CLINICAL TRIAL: NCT06662253
Title: Anti-Xa Guided Dosing of Low Molecular Weight Heparin for Prevention of Venous Thromboembolism Following Traumatic Injury: a Multicentre Pilot Randomized Trial
Acronym: PrOVE iT
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alexandre Tran (Other)
Responsible Party: Sponsor-Investigator, Alexandre Tran, Associate Scientist, Ottawa Hospital Research Institute
Organization: Ottawa Hospital Research Institute (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20240579-01H
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-09

CONDITIONS: Venous Thromboembolism (VTE); Trauma Related Injuries
Keywords: trauma; venous thromboembolism; prophylaxis
MeSH Terms: conditions — Venous Thromboembolism; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): Participants will receive Enoxaparin dosed at the discretion of the most responsible physician (MRP). In cases of severe renal insufficiency (CrCl < 30mL/min^:), the LMWH may dose reduced or changed to Heparin at the discretion of the MRP.
  Interventions: Drug: Standard of Care Dosing
- Intervention (Anti-Xa Guided) (Experimental): Participants will receive Enoxaparin 0.5 mg/kg twice daily (rounded up or down to the nearest 10 mg) the initial starting dose. Dose adjustments will be made based on trough levels drawn between the 3rd and 4th dose. The target anti-Xa level range is between 0.1 and 0.2 IU/mL. If the patient is below the target range, then the next Enoxaparin dose will be increased by 10 mg per dose with a new trough anti-Xa level 24 hours after dose modification. If the patient is above the target range, then the next Enoxaparin dose will be decreased by 10 mg per dose with a new trough anti-Xa level 24 hours after dose modification. This dose will be maintained until hospital discharge.
  Interventions: Drug: Anti-Xa Guided Dosing of Low Molecular Weight Heparin

INTERVENTIONS:
Drug: Anti-Xa Guided Dosing of Low Molecular Weight Heparin — Participants will receive Enoxaparin 0.5 mg/kg twice daily (rounded up or down to the nearest 10 mg) the initial starting dose. Dose adjustments will be made based on trough levels drawn between the 3rd and 4th dose. The target anti-Xa level range is between 0.1 and 0.2 IU/mL. If the patient is below the target range, then the next Enoxaparin dose will be increased by 10 mg per dose with a new trough anti-Xa level 24 hours after dose modification. If the patient is above the target range, then the next Enoxaparin dose will be decreased by 10 mg per dose with a new trough anti-Xa level 24 hours after dose modification. This dose will be maintained until hospital discharge.
  Arms: Intervention (Anti-Xa Guided)
Drug: Standard of Care Dosing — Participants will receive Enoxaparin dosed at the discretion of the most responsible physician (MRP). In cases of severe renal insufficiency (CrCl < 30mL/min^:), the LMWH may dose reduced or changed to Heparin at the discretion of the MRP.
  Arms: Standard of Care

SUMMARY:
This multicentre pilot trial will assess the feasibility of a full-scale, randomized trial to determine whether bloodwork guided dosing of blood thinners reduces the risk of clotting in high-risk trauma patients. Patients will receive either standard of care dosing or dosing with adjustments based on bloodwork to achieve a minimum therapeutic threshold.

DETAILED DESCRIPTION:
This multicentre pilot trial will assess the feasibility of a full-scale, randomized trial to determine whether anti-Xa guided dosing of low molecular heparin (LMWH) reduces the risk of venous thromboembolism (VTE) in high-risk trauma patients. Patients will receive either standard of care fixed dosing of Enoxaparin or 0.5 mg/kg twice daily with dose adjustments to achieve an anti-Xa trough level between 0.1 and 0.2 IU/mL.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older admitted to a hospital ward or intensive care unit following a traumatic injury involving two or more body systems (head, chest, abdomen, pelvis, extremity) and meeting at least one of the following high-risk criteria previously identified in a recent systematic review (1): age ≥ 65, body mass index ≥ 30 kg/m2, injury severity score ≥ 16, pelvic injury with activity restrictions, lower extremity injury with activity restrictions, or surgery during the index hospitalization.

To be eligible, patients must be deemed appropriate for pharmacologic prophylaxis by the most responsible physician and randomized with the intention to receive prophylaxis within 48 hours of admission. Prior to randomization, there is no restriction on whether or not patients have previously received pharmacologic or mechanical prophylaxis.

Exclusion Criteria:

1. Greater than 7 days since time of injury.
2. Requirement for therapeutic anticoagulation or dual-antiplatelet therapy
3. Unable or unwilling to receive pharmacologic prophylaxis within 48 hours of admission.
4. History of allergic reaction or sensitivity to LMWH.
5. Thrombocytopenia with platelets < 30.
6. Expected discharge or transfer from hospital within 72 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Recruitment (Patients per site per month) | Participants per site per month x 15 months
  The pilot trial will have an expected duration of 15 months during which time we hope to enroll at least 150 participants total across all sites - therefore, 5 patients/site/month. There are no maximum enrollment targets for each site.

SECONDARY OUTCOMES:
Eligibility rate | 15 months
  Proportion of screened patients who are eligible
Consent rate | 15 months
  Proportion of eligible patients who provide consent
Retention rate | 15 months
  Proportion of participants retained at follow-up
Study completion rate | 15 months
  Proportion of participants who completed all study procedures
Adherence rate | 15 months
  Adherence to study drug measured by proportion of prophylaxis doses received.
Adherence to monitoring | 15 months
  Proportion of patients with anti-Xa tests ordered appropriately
Adherence to dose adjustment | 15 months
  Proportion of doses adjusted appropriately for anti-Xa level
Adherence to anti-Xa target | 15 months
  Proportion of patients who achieved target anti-Xa range
Reasons for declining participation | 15 months
  Reasons for declining participation

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Tran, MD, MSc, FRCSC, Principal Investigator — Ottawa Hospital Research Institute; Marc Carrier, MD, MSc, FRCPC, Principal Investigator — Ottawa Hospital Research Institute